CLINICAL TRIAL: NCT00708838
Title: VLA-1 Receptors on Peripheral T Cells in Ischemic Heart Disease Patients
Brief Title: Levels of Circulating T Cells Expressing VLA-1 Collagen Receptors
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Arik Asman, Sheba Medical Center, Heart Institute
Other Study IDs: SHEBA-02-2707-AA-CTIL
Record Dates: First submitted 2008-07-01; First posted 2008-07-02 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-07

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples isolated from patients included in the study and anallysed by FACS
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1
- 2
- 3
- 4
- 5

SUMMARY:
The examination of the percentage of peripheral T cells carrying VLA-1 in ischemic heart disease patients. The hypothesis is that the percentage levels of cells carrying this integrin rise according to the severity of the ischemic heart disease.

DETAILED DESCRIPTION:
Atherosclerosis is considered an inflammatory disease in which lymphocytes have an important role. The study was disigned to find out the changes in T cell levels carrying VLA-1 involvement in this process.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of acute MI for group 1
* clinical diagnosis of ACSl for group 2
* clinical diagnosis of Chronic Heart Disease for groups 3 and 4
* Chest pain but normal heart scan for group 5

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2002-01; Primary Completion 2006-01 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The differance in percentage of T cells in the 5 different groups involved. | 2002-2006